CLINICAL TRIAL: NCT05215678
Title: Generalizability of Overweight Patients With Knee Osteoarthritis Awaiting Knee Surgery Accepting to Join a Weight Loss Randomized Trial: Protocol for a Cross-sectional Study Comparing Baseline Characteristics and Propensity of Patients Accepting/Declining Enrolment
Brief Title: Characteristics of Patients Declining INKA Trial Participation
Acronym: n-INKA
Status: Completed | Type: Observational
Sponsor: Marius Henriksen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Other Study IDs: N-INKA
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- INKA participants: Individuals eligible and accepting participation in the INKA trial (NCT05172843)
  Interventions: Other: Acceptance of invitation to trial participation
- n-INKA participants: Individuals eligible and declining participation in the INKA trial (NCT05172843)
  Interventions: Other: Declining invitation to trial participation

INTERVENTIONS:
Other: Acceptance of invitation to trial participation — Individuals who are eligible for and accept participation in the INKA trial (NCT05172843)
  Groups: INKA participants
Other: Declining invitation to trial participation — Individuals who are eligible for participation in the INKA trial (NCT05172843) but decline the invitation to participate
  Groups: n-INKA participants

SUMMARY:
The objective of this study is to compare baseline characteristics of overweight knee OA patients accepting vs. declining enrolment in the INKA trial (NCT05172843) to explore if enrolled patients differ systematically from the declining participants with respect to both measured as well as unmeasured baseline characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or more
2. A clinical and radiological diagnosis of knee OA
3. BMI ≥ 30 kg/m2
4. Motivated for weight loss as by the provided program
5. Signed informed consent.

Exclusion Criteria:

1. The scheduled surgery is for revision of an existing prosthesis
2. Planned surgery for more than one knee within the observation period
3. KA indication due to sequelae of fracture(s)
4. Injection of medication or substances in the target knee within 3 months prior to participation
5. Immuno-inflammatory arthritis as cause of the knee OA
6. Current systemic treatment with glucocorticoids equivalent to > 7.5 mg of prednisolone/day
7. Previous or planned obesity surgery
8. Inability to understand or read Danish incl. instructions and questionnaires
9. Any other condition or impairment that, in the opinion of the investigator (or his/her delegate), makes a potential participant unsuitable for participation or which obstruct participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients found eligible in INKA study (inclusion criteria for INKA (NCT05172843) and accepting and declining enrolment in the INKA study are invited to participate in our study.
  Study participants will be adults (i.e. at least 18 years old), have a diagnosis of knee osteoarthritis with an indication for primary knee arthroplasty (unicondylar or total arthroplasty), and be obese (BMI≥30 kg/m2).
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Oxford knee score | Baseline
  The Oxford Knee Score (OKS) is a 12-item Patient Reported Outcome questionnaire developed specifically to assess the patient's perspective on the outcomes of knee arthroplasty (KA) with respect to combined pain and physical function. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. Thus, a total score is calculated that ranges from 0 and 48, with 48 indicating the best outcome.

SECONDARY OUTCOMES:
Health outcome and quality of life survey (EQ-5D-5L) | Baseline
  EQ-5D-5L is a standardized patient-reported instrument for use as a measure of health outcome and quality of life. EQ-5D-5L is designed for self-completion by respondents and is ideally suited for use in surveys.
  The EQ-5D-5L consists of a descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 1 to 3. It is simple, taking only a few minutes to complete. Instructions to respondents are included in the questionnaire.
  The EQ-5D VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'.
Analgesic use | Baseline
  At clinical outcome assessment visit, the participants will be interviewed by an investigator about their use of analgesics since last visit. The interview will be focused on intake of
  1. Paracetamol/acetaminophen
  2. NSAIDS
  3. Acetylic acids
  4. Opioids The use of these analgesics will be recorded as a 0-3 points Likert scale (0, never; 1, rarely; 2, 2-3 times per week; 3, daily or almost daily).
The Knee Injury and Osteoarthritis Outcome Score - 12 item short form (KOOS-12) | Baseline
  KOOS-12 provides scale scores for knee-specific Pain, Function and QOL, along with a summary measure of overall knee impact.
  Each item is scored from 0 to 4, with 0 representing no knee problems and 4 representing extreme knee problems. The separate KOOS-12 Pain, Function and QOL scale scores are calculated, in which item responses are summed.
  The KOOS-12 Summary knee impact score is calculated as the average of the KOOS-12 Pain, KOOS-12 Function and KOOS-12 QOL scale scores. A Summary impact score is not calculated if any of the three scale scores are missing. The KOOS-12 Summary impact score also ranges from 0 to 100, where 0 is the worst possible and 100 is the best possible score.
Patient's global assessment of impact of the knee in daily life (PGA) | Baseline
  The participant's assessment of the impact of their knee on everyday life is measured as the response to the question "Taking into account all the activities you have during your daily life, your level of pain, and your functional impairment, how much does your [left/right] knee impact your daily life?". A 100 mm visual analogue scale (VAS) will be used as assessment instrument with anchors: 0 = "No impact" and 100 = "Worst imaginable impact".
Body weight | Baseline
  The participants body weight is transferred from the medical records of their visit in the orthopaedic outpatient clinic.
Brief Illness perception questionnaire (B-IPQ) | Baseline
  B-IPQ is a generic 9-item questionnaire developed to rapidly assess the cognitive and emotional representations in a variety of illnesses. B-IPQ is a short version of the 84-item revised illness perception questionnaire (IPQ-R) (21). B-IPQ assesses perceptions on the following five dimensions: Identity, Cause, Timeline, Consequences and Cure-Control. Five of the items assess cognitive illness representations; two of the items assess emotional representations; and one item assesses illness comprehensibility. The 8 items are scored on a 0-3 Likert scale with descriptors (none or extreme) at either end.

CONTACTS AND LOCATIONS:
Overall Officials: Søren Overgaard, DMSc, Study Chair — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- The Parker Institute, Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Decision to share IPD with other researchers will be made at a later stage, including criteria for sharing.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-09): https://cdn.clinicaltrials.gov/large-docs/78/NCT05215678/Prot_SAP_000.pdf